CLINICAL TRIAL: NCT00248287
Title: Randomized Phase II Study of Weekly Irinotecan/Carboplatin (ICb) With or Without Cetuximab (Erbitux) in Patients With Metastatic Breast Cancer
Brief Title: PhII ICb With/Without Erbitux in MBC Pts
Acronym: CA225200
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Bristol-Myers Squibb (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04070; CA225200 (Other: Bristol-Myers-Squibb)
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Irinotecan; Carboplatin; Cetuximab

ARMS (2):
- Arm 1 (Active Comparator): irinotecan 90 mg/m2 and carboplatin AUC=2.0 on Days 1 and 8 of each 21-day cycle (Arm 1, ICb)
  Interventions: Drug: Irinotecan + Carboplatin
- Arm 2 (Experimental): irinotecan 90mg/m2, carboplatin AUC=2.0 on Days 1 and 8 of each 21- day cycle plus Erbitux 400 mg/m2 Week 1 and then 250 mg/m2 weekly thereafter, (Arm 2, ICb+Erbitux)
  Interventions: Drug: irinotecan + Carboplatin + erbitux

INTERVENTIONS:
Drug: Irinotecan + Carboplatin — irinotecan 90 mg/m2 and carboplatin AUC=2.0 on Days 1 and 8 of each 21-day cycle
  Arms: Arm 1
Drug: irinotecan + Carboplatin + erbitux — irinotecan 90mg/m2, carboplatin AUC=2.0 on Days 1 and 8 of each 21- day cycle plus Erbitux 400 mg/m2
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine the objective response rates produced by irinotecan and carboplatin therapy with or without Erbitux in patients with Metastatic Breast Cancer.

ELIGIBILITY:
INCLUSION CRITERIA:

Male and female patients will be eligible for inclusion in this study if they meet all of the following criteria:

* Has cytologically or pathologically confirmed, breast cancer with documented HER2+ (positive) (3+ by IHC or FISH+) or HER2- (negative) disease. ER, PR, and HER2 status must be documented in the electronic Case Report Form (eCRF) NOTE: Patients whose breast cancers are HER2 (2+) by IHC must undergo FISH testing to confirm HER2+ (positive) status.
* Has clinically confirmed Stage IV metastatic breast cancer (MBC)
* Has undergone prior Herceptin therapy if breast cancer is HER2+ (positive)
* Has measurable MBC as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria

NOTE: Ascites, pleural effusion, and bone metastases are not considered measurable.

* Has had up to 1 prior chemotherapy regimens for metastatic disease. Previously untreated disease is permitted.
* Has had no prior treatment with irinotecan, carboplatin, or cisplatin
* Has an ECOG Performance Status (PS) 0-2
* Is greater than 18 years of age
* Please see protocol for specific details regarding appropriate laboratory values for inclusion to the study.
* Any prior radiation therapy has been completed > 2 weeks prior to the start of study treatment

NOTE: Previously irradiated lesions will not be evaluable; however, these patients will still be eligible. Patients must have at least 1 measurable lesion at baseline.

* Has had a negative serum pregnancy test within 7 days prior to registration (female patients of childbearing potential). A pregnancy test is also required within 7 days of Dose 1.
* If fertile, patient (male or female) has agreed to use an acceptable method of birth control to avoid pregnancy for the duration of the study and for a period of 6 months thereafter.
* Has signed a Patient Informed Consent Form
* Has signed a Patient Authorization Form (HIPAA)
* Has paraffin-embedded breast cancer tissue (either paraffin blocks or 20 unstained slides) available for analysis of EGFR, cytokeratin, and other biological markers. These samples will be sent to the Molecular Profiling Institute (MPI; see Appendix VII).

NOTE: Availability of samples should be confirmed prior to randomization (at latest, prior to first dose).

EXCLUSION CRITERIA:

* Has Stage I-III breast cancer or nonmeasurable metastatic breast cancer, or any disease other than that described in inclusion criterion #1
* Has received prior treatment with irinotecan, carboplatin, or cisplatin
* Is receiving any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s)
* Has received prior therapy which specifically and directly targets the EGFR pathway. Prior Herceptin is required for HER2+ patients.
* Has had prior severe infusion reaction to a monoclonal antibody
* Has received organ allograft(s) other than corneal, bone, or skin
* Has clinically significant uncontrolled cardiac disease (eg, congestive heart failure, symptomatic coronary artery disease or cardiac arrhythmias not well-controlled with medication) or has had a myocardial infarction < 12 months
* Has ongoing peripheral neuropathy > Grade I
* Has evidence of symptomatic or untreated central nervous system (CNS) metastases (unless CNS metastases have been irradiated). Chronic steroid treatment for the treatment of CNS metastases must have been discontinued for greater than 4 weeks prior to study enrollment.
* Has any other significant comorbidity that, in the opinion of the clinical investigator, might compromise any aspect of the study
* Has active or uncontrolled infection
* Has acute hepatitis or is known to be HIV positive
* Has a history of other malignancy within the last 5 years which could affect the diagnosis or assessment of MBC, with the exception of carcinoma of the cervix in situ, carcinoma of the bladder in situ, and basal cell carcinoma
* Has previously completed a chemotherapy regimen within 3 weeks prior to the start of study treatment, or has related toxicities unresolved prior to the start of study treatment

NOTE: If patient was receiving prior weekly or daily chemotherapy, he/she may begin study therapy 2 weeks after stopping prior therapy provided all toxicities have resolved; peripheral neuropathy must be less than Grade I as per exclusion criterion #8 above.

* Has had major surgery within 3 weeks from the start of study treatment, without complete recovery
* Has participated in any investigational drug study within 4 weeks preceding the start of study treatment
* Has received a concurrent immunotherapy or hormonal anticancer agent within 2 weeks prior to the start of the study treatment
* Is receiving a tyrosine kinase inhibitor (ie, IressaTM)
* Has had any prior stem cell or bone marrow transplant for any prior hematologic malignancy
* Is pregnant or lactating
* Is unable to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2005-07-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A. O'Shaughnessy, MD, Principal Investigator — US Oncology Research
Locations (58):
- United States (58):
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Hematology Oncology Asscociates, Phoenix, Arizona
  - Northern AZ Hematology & Oncology Assoc, Sedona, Arizona
  - Rocky Mountain Cancer Center-Rose, Denver, Colorado
  - Northwestern Connecticut Oncology Hematology Associates, Torrington, Connecticut
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Hematology Oncology Associates of IL, Chicago, Illinois
  - Central Indiana Cancer Center, Indianapolis, Indiana
  - Kansas City Cancer-Southwest, Overland Park, Kansas
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Arch Medical Services, Inc, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - NH Oncology-Hematology PA, Hooksett, New Hampshire
  - Hematology-Oncology Associates of NNJ, P.A., Morristown, New Jersey
  - Summit Medical Group, Summit, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - New York Oncology Hematology, PC, Rexford, New York
  - Interlakes Oncology Hematology, PC, Rochester, New York
  - Raleigh Hematology Oncology Clinic, Cary, North Carolina
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Cancer Center of the Carolinas, Seneca, Seneca, South Carolina
  - Texas Cancer Center-Abilene(South), Abilene, Texas
  - Texas Cancer Center, Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology, P.A. - Bedford, Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - The Texas Cancer Center, Dallas, Texas
  - Texas Oncology Center - Denton, Denton, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - San Antonio Tumor & Blood Clinic, Fredericksburg, Texas
  - Texas Oncology, P.A., Houston, Texas
  - Longview Cancer Center, Longview, Texas
  - South Texas Cancer Center-McAllen, McAllen, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - HOAST - New Braunfels, New Braunfels, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center-Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Waco Cancer Care and Research Center, Waco, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onc and Hem Associates of SW VA, Inc., Salem, Virginia
  - Puget Sound Cancer Center-Emonds, Edmonds, Washington
  - Puget Sound Cancer Center-Seattle, Seattle, Washington
  - Cancer Care Northwest-South, Spokane, Washington
  - Northwest Cancer Specialists-Vancouver, Vancouver, Washington
  - Yakima Valley Mem Hosp/North Star Lodge, Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Irinotecan+Carboplatin: Patients treated with Irinotecan + Carboplatin
- Irinotecan+Carboplatin+Cetuximab: Patients treated with Irinotecan + Carboplatin + Cetuximab
Period: Overall Study
Arm/Group | Irinotecan+Carboplatin | Irinotecan+Carboplatin+Cetuximab
Started | 75 | 79
Completed | 51 | 60
Not Completed | 24 | 19
Not completed — Adverse Event | 11 | 10
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Investigator Request | 4 | 3
Not completed — Patient Request | 5 | 3
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Irinotecan+Carboplatin | Irinotecan+Carboplatin+Cetuximab | Total
Number analyzed (Participants) | 75 | 79 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.4) | 54.9 (10.7) | 54.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 79 | 154
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 59 | 69 | 128
  Black | 14 | 8 | 22
  Hispanic | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 75 | 79 | 154

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rates (ORR)
Description: To determine the objective response rates (CR + PR). Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: 2 years
Population: Evaluable population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Irinotecan+Carboplatin | Irinotecan+Carboplatin+Cetuximab
Number analyzed (Participants) | 66 | 71
Percentage of Participants | 36.4 [24.9 to 49.1] | 36.6 [25.5 to 48.9]

2. Secondary Outcome: Duration of Response
Description: The duration of response is measured from the time measurement criteria are first met for CR/PR until the first date that recurrent or progressive disease is objectively documented.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: From date of randomization until the date of first documented progression or the date of death from any cause, whichever came first, assessed up to 60 months.
Population: For patients who achieve a major objective response (CR or PR) the time to response will be assessed as the date of registration to the date of response.
Measure: Median (Full Range); unit: months
Arm/Group | Irinotecan+Carboplatin | Irinotecan+Carboplatin+Cetuximab
Number analyzed (Participants) | 24 | 26
months | 5.4 [2.0 to 34.3] | 6.0 [1.4 to 41.3]

3. Secondary Outcome: Median Time of Progression-free Survival (PFS)
Description: PFS is measured from the date of randomization to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at last contact date.
Time Frame: 2 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan+Carboplatin | Irinotecan+Carboplatin+Cetuximab
Number analyzed (Participants) | 75 | 79
months | 4.4 [3.2 to 5.8] | 4.6 [3.5 to 5.5]

4. Secondary Outcome: Median Overall Survival (OS)
Description: OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: 2 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan+Carboplatin | Irinotecan+Carboplatin+Cetuximab
Number analyzed (Participants) | 75 | 79
months | 12.5 [10.6 to 17.1] | 14.6 [10.4 to 16.9]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treated patients only, assessed at each treatment visit.
Arm/Group | Irinotecan+Carboplatin | Irinotecan+Carboplatin+Cetuximab
All-Cause Mortality (participants affected / at risk) | 1/75 | 0/79
Serious Adverse Events (participants affected / at risk) | 14/75 | 18/79
Other Adverse Events (participants affected / at risk) | 73/75 | 79/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan+Carboplatin (N=75) | Irinotecan+Carboplatin+Cetuximab (N=79)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ALLERGIC REACTION (Immune system disorders) | 1 (1) | 0 (0)
ANAPHYLAXIS (Immune system disorders) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
BACTERIAL RESISTANCE (Infections and infestations) | 1 (1) | 0 (0)
CONFUSION (General disorders) | 1 (1) | 0 (0)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 8 (8) | 6 (6)
DIARRHEA (Gastrointestinal disorders) | 5 (5) | 9 (10)
EMBOLISM PULMONARY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
FEVER (General disorders) | 1 (1) | 0 (0)
HYPERBILIRUBINEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERSENSITIVITY REACTION (NOS) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
INFECTION UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2)
NAUSEA AND VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
REACTION INJECTION SITE (NOS) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 2 (2)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
WEAKNESS GENERALIZED (General disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan+Carboplatin (N=75) | Irinotecan+Carboplatin+Cetuximab (N=79)
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 (13) | 19 (30)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
ALLERGIC REACTION (Immune system disorders) | 1 (1) | 5 (7)
ALOPECIA (Skin and subcutaneous tissue disorders) | 20 (23) | 27 (29)
ANEMIA (Blood and lymphatic system disorders) | 47 (189) | 40 (132)
ANOREXIA (Gastrointestinal disorders) | 18 (23) | 19 (23)
AST INCREASED (Metabolism and nutrition disorders) | 2 (4) | 6 (9)
CONSTIPATION (Gastrointestinal disorders) | 15 (20) | 11 (11)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (9)
DEHYDRATION (Gastrointestinal disorders) | 9 (9) | 14 (20)
DIARRHEA (Gastrointestinal disorders) | 50 (91) | 58 (130)
DIZZINESS (Nervous system disorders) | 6 (7) | 9 (16)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (4) | 19 (20)
EDEMA (Blood and lymphatic system disorders) | 2 (3) | 4 (6)
FATIGUE (General disorders) | 45 (105) | 51 (110)
FEVER (General disorders) | 9 (10) | 2 (2)
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 10 (12) | 11 (13)
HEADACHE (General disorders) | 2 (2) | 6 (8)
HOT FLASHES (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 10 (14) | 14 (26)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 11 (30) | 22 (43)
HYPOTENSION (Vascular disorders) | 4 (4) | 2 (2)
LEUCOPENIA (Blood and lymphatic system disorders) | 29 (177) | 32 (170)
LYMPHOPENIA (Blood and lymphatic system disorders) | 5 (39) | 5 (24)
MUCOSITIS (Infections and infestations) | 7 (8) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (12) | 4 (7)
NAUSEA (Gastrointestinal disorders) | 55 (102) | 47 (90)
NEUROPATHY (Nervous system disorders) | 6 (17) | 8 (11)
NEUTROPENIA (Blood and lymphatic system disorders) | 53 (242) | 56 (257)
PAIN (General disorders) | 6 (7) | 3 (3)
PARESTHESIA (Nervous system disorders) | 2 (2) | 4 (4)
PHOSPHATASE ALKALINE INCREASED (Metabolism and nutrition disorders) | 2 (3) | 4 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6)
RASH (Skin and subcutaneous tissue disorders) | 14 (22) | 56 (105)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (7)
STOMATITIS (Gastrointestinal disorders) | 3 (3) | 5 (6)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 39 (138) | 32 (90)
VOMITING (Gastrointestinal disorders) | 30 (38) | 34 (50)
WEAKNESS (General disorders) | 4 (7) | 10 (14)
WEIGHT LOSS (General disorders) | 4 (5) | 12 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-04-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT00248287/Prot_SAP_000.pdf